CLINICAL TRIAL: NCT06254586
Title: Effects of Blood Flow Restriction Training on Heart Rate, Blood Pressure, Mean Arterial Pressure, and Limb Girth During Resisted Exercises Versus Aerobic Exercise in Healthy Individuals.
Brief Title: Effects of Blood Flow Restriction Training on Exercises in Healthy Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THIAGU 01
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Health, Subjective
Keywords: Blood flow Restriction Training; Blood Pressure; Heart Rate; Mean Arterial Pressure; Muscle Girth
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): This group received a single session of low-intensity cycling for 20 minutes.
  Interventions: Procedure: Aerobic exercises
- Resisted exercises (Active Comparator): This group received four sets of 15 repetitions of knee extension, hamstring curls, and standing calf raises (20-40% 1RM) with a 30 sec to 1 minute rest period between sets.
  Interventions: Procedure: Resisted exercises

INTERVENTIONS:
Procedure: Aerobic exercises — This group received a single session of low-intensity cycling for 20 minutes. A period of reperfusion (3 to 5 minutes) were provided in both groups after 10 minutes of exercise training by deflating the BFR cuffs. The cuffs were inflated after 5 minutes of reperfusion, and the exercises were completed in both groups.
  Arms: Aerobic exercise
Procedure: Resisted exercises — This group received four sets of 15 repetitions of knee extension, hamstring curls, and standing calf raises (20-40% 1RM) with 30 sec to 1 minute rest period between sets. A period of reperfusion (3 to 5 minutes) were provided in both groups after 10 minutes of exercise training by deflating the BFR cuffs. The cuffs were inflated after 5 minutes of reperfusion, and the exercises were completed in both groups.
  Arms: Resisted exercises

SUMMARY:
Partial restriction of blood flow to working muscles during exercise is proven to increase muscle mass and strength even with low-intensity of exercise. Blood Flow Restriction Training (BFRT) is also beneficial to improve the maximum rate of oxygen consumption (VO2max), bone health, and vascular health. Recent studies focus on its effects beyond the musculoskeletal system. Post-exercise hypotension is a known acute physiological response that happens after intense exercise. Early studies demonstrated BFRT might amplify the acute hypotensive effects with low intensity of exercise. However, it's not clear what type of exercise would help to lower blood pressure when it is combined with BFRT.

DETAILED DESCRIPTION:
Partial restriction of blood flow to working muscles during exercise is proven to increase muscle mass and strength even with low-intensity of exercise. Blood Flow Restriction Training (BFRT) is also beneficial to improve the maximum rate of oxygen consumption (VO2max), bone health, and vascular health. Recent studies focus on its effects beyond the musculoskeletal system. Post-exercise hypotension is a known acute physiological response that happens after intense exercise. Early studies demonstrated BFRT might amplify the acute hypotensive effects with low intensity of exercise. However, it's not clear what type of exercise would help to lower blood pressure when it is combined with BFRT. Considering BFRT, it's safe to implement among hypertensive individuals as per recent studies. It's still unclear what type of exercise would benefit maximum in reducing blood pressure while using it along BFR. The study aims to determine whether BFRT can influence BP, MAP, HR, and muscle girth differently while doing resisted exercises and aerobic exercise. Understanding the effects of BFRT on these parameters can provide valuable insights for optimizing exercise protocols and improving overall health outcomes. In general, this study can also add to the increasing amount of studies about the possible advantages and drawbacks of BFRT, and provide guidance on how to design exercise programs for people with borderline hypertension or in those with early phase of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of both gender, between the ages of 18 and 35 years
* Adults who are not participating in any regular exercise/fitness programmes for the last three months

Exclusion Criteria:

* Adults with previous history of cardiovascular diseases, or with pathological changes in ECG
* Adults with concomitant illness such as diabetes, hypertension, or kidney diseases
* Chronic smokers or alcoholics
* Those with recent history of injury to lower limbs or with implants in lower limbs

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | Baseline
  The chest strap heart rate monitors can continuously monitor heart rate throughout the day. These devices use optical sensors or electrodes to detect changes in blood flow and provide real-time data.
Heart rate | After 1 minute
  The chest strap heart rate monitors can continuously monitor heart rate throughout the day. These devices use optical sensors or electrodes to detect changes in blood flow and provide real-time data.
Heart rate | After 3 minutes
  The chest strap heart rate monitors can continuously monitor heart rate throughout the day. These devices use optical sensors or electrodes to detect changes in blood flow and provide real-time data.
Heart rate | After 5 minutes
  The chest strap heart rate monitors can continuously monitor heart rate throughout the day. These devices use optical sensors or electrodes to detect changes in blood flow and provide real-time data.
Heart rate | After 15 minutes
  The chest strap heart rate monitors can continuously monitor heart rate throughout the day. These devices use optical sensors or electrodes to detect changes in blood flow and provide real-time data.
Heart rate | After 30 minutes
  The chest strap heart rate monitors can continuously monitor heart rate throughout the day. These devices use optical sensors or electrodes to detect changes in blood flow and provide real-time data.
Blood pressure | Baseline
  BP monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Blood pressure | After 1 minute
  BP monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Blood pressure | After 3 minutes
  BP monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Blood pressure | After 5 minutes
  BP monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Blood pressure | After 15 minutes
  BP monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Blood pressure | After 30 minutes
  BP monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Mean arterial pressure | Baseline
  Mean arterial pressure monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Mean arterial pressure | After 1 minute
  Mean arterial pressure monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Mean arterial pressure | After 3 minutes
  Mean arterial pressure monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Mean arterial pressure | After 5 minutes
  Mean arterial pressure monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Mean arterial pressure | After 15 minutes
  Mean arterial pressure monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Mean arterial pressure | After 30 minutes
  Mean arterial pressure monitor devices use an inflatable cuff to measure blood pressure and detect pulsations to determine the heart rate.
Muscle girth | Baseline
  For biceps measurement, the individual should flex their arm at a 90-degree angle.
  Place the tape measure around the midpoint of the upper arm, making sure it is snug but not tight.
  Record the measurement in inches or centimeters.
Muscle girth | After 1 minute
  For biceps measurement, the individual should flex their arm at a 90-degree angle.
  Place the tape measure around the midpoint of the upper arm, making sure it is snug but not tight.
  Record the measurement in inches or centimeters.
Muscle girth | After 3 minutes
  For biceps measurement, the individual should flex their arm at a 90-degree angle.
  Place the tape measure around the midpoint of the upper arm, making sure it is snug but not tight.
  Record the measurement in inches or centimeters.
Muscle girth | After 5 minutes
  For biceps measurement, the individual should flex their arm at a 90-degree angle.
  Place the tape measure around the midpoint of the upper arm, making sure it is snug but not tight.
  Record the measurement in inches or centimeters.
Muscle girth | After 15 minutes
  For biceps measurement, the individual should flex their arm at a 90-degree angle.
  Place the tape measure around the midpoint of the upper arm, making sure it is snug but not tight.
  Record the measurement in inches or centimeters.
Muscle girth | After 30 minutes
  For biceps measurement, the individual should flex their arm at a 90-degree angle.
  Place the tape measure around the midpoint of the upper arm, making sure it is snug but not tight.
  Record the measurement in inches or centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Nambi, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No